CLINICAL TRIAL: NCT06820073
Title: Effects of an Intervention with Global Postural Reeducation (GPR) Using the K-Stretch Hammock on Posture, Functionality, and Musculoskeletal Discomfort in the Cervical and Lumbar Regions of Technical and Administrative Staff At San Jorge University
Brief Title: Effects of GPR with K-Stretch Hammock on Posture and Musculoskeletal Discomfort
Acronym: GPR-KS_PI24/47
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad San Jorge (Other)
Responsible Party: Principal Investigator, Cristina Comeras, Principal Investigator, Universidad San Jorge
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: GPR-KS
Record Dates: First submitted 2025-01-15; First posted 2025-02-11 (Actual); Last update posted 2025-02-11 (Actual); Status verified 2025-02

CONDITIONS: Cervical and Lumbar Musculoskeletal Discomfort
Keywords: musculoskeletal discomfort; Lumbar discomfort; Cervical discomfort; Global Postural Reeducation (RPG); K-Stretch hammock; Workplace intervention; Posture improvement; Quality of life enhancement

STUDY DESIGN:
Intervention Model Description: This study employs an interventional, two-group, randomized, controlled design to evaluate the effects of Global Postural Reeducation (RPG) using the K-Stretch hammock on musculoskeletal discomfort and related outcomes. Participants are randomly assigned to either Group 1, which undergoes the intervention in the first six weeks, or Group 2, which receives the same intervention after Group 1 completes its post-intervention assessment. Each group participates in 12 sessions, lasting 30 minutes each, conducted twice weekly. The intervention involves targeted stretching techniques focused on improving posture, reducing musculoskeletal discomfort, and enhancing flexibility and alignment. Assessments are conducted at baseline, after Group 1 intervention, and after Group 2 intervention to compare pre- and post-intervention outcomes and ensure a robust evaluation of the intervention's effectiveness.
Who Masked: Investigator, Outcomes Assessor
Masking Description: This study is open-label, and no masking is applied. Both participants and investigators are aware of the group assignments and the intervention being conducted. However, data analysis is performed on pseudonymized datasets to maintain objectivity and confidentiality. The individual responsible for assigning participant codes is not involved in data analysis, ensuring that any potential bias is minimized during the statistical evaluation process.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Immediate Intervention Group: Participants receive the RPG intervention using the K-Stretch hammock (Experimental): Participants in this arm will begin the intervention immediately after enrollment. The intervention involves 12 sessions of Global Postural Reeducation (RPG) using the K-Stretch hammock, delivered over six weeks with two 30-minute sessions per week. These sessions aim to improve posture, reduce cervical and lumbar musculoskeletal discomfort, and enhance flexibility and alignment.
  Participants will undergo assessments before and after the intervention to measure changes in musculoskeletal discomfort, functional capacity, range of motion, muscle tone, stress levels, and quality of life. This arm serves to evaluate the immediate effects of the RPG intervention, providing data for comparison with the delayed intervention group.
  Interventions: Behavioral: Global Postural Reeducation (RPG) using the K-Stretch hammock
- Delayed Intervention Group: Participants receive the RPG intervention after Group 1 completes it. (Experimental): Participants in this arm will receive the Global Postural Reeducation (RPG) intervention using the K-Stretch hammock after Group 1 completes their intervention and post-intervention assessments. The intervention consists of 12 sessions conducted over six weeks, with two 30-minute sessions per week.
  The sessions are designed to improve posture, reduce cervical and lumbar musculoskeletal discomfort, and enhance flexibility and alignment. Assessments for this group will include a baseline evaluation, conducted prior to the delayed intervention period, and a post-intervention assessment to measure changes in musculoskeletal discomfort, functional capacity, range of motion, muscle tone, stress levels, and quality of life.
  This arm allows for a comparative analysis of immediate versus delayed intervention outcomes to assess the overall effectiveness of the RPG program.
  Interventions: Behavioral: Global Postural Reeducation (RPG) using the K-Stretch hammock

INTERVENTIONS:
Behavioral: Global Postural Reeducation (RPG) using the K-Stretch hammock — The intervention involves Global Postural Reeducation (RPG) using the K-Stretch hammock. This therapeutic approach focuses on sustained stretching of muscle chains to improve posture, reduce cervical and lumbar musculoskeletal discomfort, and enhance flexibility. Participants complete 12 sessions over six weeks, with two 30-minute sessions per week. Each session includes guided exercises that target muscle imbalances, improve alignment, and alleviate tension caused by prolonged sedentary behavior. The K-Stretch hammock provides support for optimized stretching and alignment during the exercises.

SUMMARY:
This study aims to evaluate the effects of Global Postural Reeducation (RPG) using the K-Stretch hammock on workers at San Jorge University who experience neck and lower back discomfort due to prolonged sitting. The primary goal is to examine how this intervention impacts posture, musculoskeletal discomfort, flexibility, and range of motion, as well as participants' quality of life, stress levels, and sleep quality.

Neck and lower back discomfort are common issues that significantly impact individuals' quality of life and work performance. Global Postural Reeducation (RPG) is a therapeutic approach that focuses on stretching and strengthening muscle chains to improve posture and alleviate discomfort. This study is innovative in applying RPG combined with a specialized K-Stretch hammock to assess its potential benefits in a workplace setting.

Participants will include 32 administrative staff members aged 19 to 65 who work predominantly in seated positions and meet specific inclusion criteria. They will undergo a 6-week program involving bi-weekly 30-minute sessions. The study will also compare pre- and post-intervention results to evaluate changes in musculoskeletal discomfort, functional abilities, and physical alignment. Findings from this study may contribute to developing effective workplace interventions for musculoskeletal health.

DETAILED DESCRIPTION:
Here is the revised version of your text without dashes, bullet points, or special characters:

This clinical trial investigates the effects of Global Postural Reeducation combined with the use of a specialized K-Stretch hammock on improving musculoskeletal discomfort and related physical and psychosocial outcomes in a workplace setting. The study specifically targets neck and lumbar musculoskeletal discomfort among technical and administrative staff at San Jorge University who are exposed to prolonged sedentary work conditions.

The research is designed as a two-group randomized controlled intervention study focusing on the application of a structured RPG program. Participants are randomized into two groups: the intervention group, referred to as Group 1, and a delayed-intervention group, referred to as Group 2. Group 1 undergoes the RPG intervention during the initial six-week phase, while Group 2 receives the same intervention after the post-intervention evaluation of Group 1.

The RPG methodology utilizes sustained muscle chain stretches facilitated by the K-Stretch hammock, which supports participants in achieving better posture and reducing tension in key areas prone to discomfort due to sedentary behavior. The intervention includes twelve sessions, each lasting thirty minutes, conducted twice weekly. Sessions emphasize targeted stretching techniques for muscle chains affecting the cervical and lumbar spine, integrating relaxation and alignment strategies to promote improved physical and mental well-being.

Key features of the protocol include several aspects. The study type is interventional. Allocation is randomized. The intervention model is sequential assignment. Masking is not applied in this open-label trial. The primary purpose is treatment.

The objectives of the study are as follows. The trial seeks to evaluate the impact of RPG with K-Stretch on musculoskeletal discomfort in cervical and lumbar regions. It aims to assess improvements in flexibility, range of motion, and postural alignment. Additionally, it investigates secondary outcomes, including perceived stress, sleep quality, and overall quality of life.

The intervention procedures are standardized to ensure consistency. Each session includes a warm-up phase with gentle preparatory stretches to enhance mobility. This is followed by a main phase consisting of targeted RPG exercises using the K-Stretch hammock to address muscle imbalances, posture correction, and tension relief. The session concludes with a cool-down phase involving relaxation techniques to consolidate benefits and minimize post-exercise discomfort.

Assessment tools and timelines are employed to measure both physical and psychosocial variables. Physical outcomes include musculoskeletal discomfort measured by the Cornell Musculoskeletal Discomfort Questionnaire, functional capacity assessed with the Oswestry Disability Index and Neck Disability Index, range of motion measured with a goniometer, muscle tone evaluated using the Myoton device, and postural assessment conducted with the Motiphysio Scanner and Spinal Mouse technology. Psychosocial outcomes include quality of life measured by the EQ-5D Questionnaire and stress levels assessed using the Perceived Stress Scale. Evaluations are conducted at baseline before the intervention, after the intervention for Group 1, and finally after the intervention for Group 2.

Data management and analysis follow strict ethical guidelines. Data are pseudonymized using unique alphanumeric codes assigned to each participant to ensure confidentiality. Statistical analysis will be conducted using software tools such as SPSS, focusing on within-group and between-group comparisons. The primary endpoint is the reduction in musculoskeletal discomfort, while secondary endpoints include functional and psychosocial improvements.

This trial is expected to provide robust evidence supporting the use of RPG with the K-Stretch hammock as a workplace intervention to mitigate musculoskeletal issues. By addressing physical and psychosocial health, the intervention may enhance productivity, reduce absenteeism, and contribute to a healthier work environment.

By integrating innovative techniques with rigorous assessment, this study aims to contribute significantly to the field of occupational health and rehabilitative practices. The findings will inform future research and practical applications for managing musculoskeletal discomfort in various populations.

ELIGIBILITY:
Inclusion Criteria:

* Be a university administrative or technical staff member over 18 years old who works in a seated position during the workday.
* Have at least one year of experience in the current position.
* Present nonspecific cervical and/or lumbar musculoskeletal discomfort.

Exclusion Criteria:

* Be pregnant or breastfeeding.
* Have a diagnosed condition that prevents participation in an RPG session using the K-Stretch hammock.
* Participate in activities involving RPG and/or back health programs.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2025-02-01 (Estimated); Primary Completion 2025-04-20 (Estimated); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
Cervical and Lumbar Musculoskeletal Discomfort | Immediate Intervention Group: Just before the intervention, immediately after (6 weeks), and 6 weeks post-intervention (12 weeks). Delayed Intervention Group: 6 weeks before the intervention, just before, and immediately after the intervention (6 weeks).
  Measured using the Cornell Musculoskeletal Discomfort Questionnaire (CMDQ). This tool assesses the severity and frequency of discomfort in cervical and lumbar regions.
Cervical and Lumbar Musculoskeletal Discomfort Scale | Immediate Intervention Group: Just before the intervention, immediately after (6 weeks), and 6 weeks post-intervention (12 weeks). Delayed Intervention Group: 6 weeks before the intervention, just before, and immediately after the intervention (6 weeks).
  Measured using a Numerical Rating Scale (NRS)
Improvement in Quality of Life | Immediate Intervention Group: Just before the intervention, immediately after (6 weeks), and 6 weeks post-intervention (12 weeks). Delayed Intervention Group: 6 weeks before the intervention, just before, and immediately after the intervention (6 weeks).
  Assessed using the EUROQOOL-5D questionnaire, which evaluates mobility, self-care, usual activities, pain or discomfort, and anxiety or depression to determine participants' overall quality of life.
  The EQ-5D-5L index value ranges from -0.285 (worst possible health state) to 1 (best possible health state), where higher scores indicate a better quality of life. Additionally, the EQ-VAS (EuroQol Visual Analogue Scale) ranges from 0 to 100, with 0 representing "the worst health state imaginable" and 100 representing "the best health state imaginable."

SECONDARY OUTCOMES:
Improvement in Functional Capacity of Low Back | Immediate Intervention Group: Just before the intervention, immediately after (6 weeks), and 6 weeks post-intervention (12 weeks). Delayed Intervention Group: 6 weeks before the intervention, just before, and immediately after the intervention (6 weeks).
  Assessed using the Oswestry Low Back Disability Questionnaire (ODI). This tool evaluates limitations in daily activities and the functional impact of lumbar discomfort.
  The score ranges from 0 to 100, where higher scores indicate greater disability:
  0-20%: Minimal disability 21-40%: Moderate disability 41-60%: Severe disability 61-80%: Crippling disability 81-100%: Patient is either bed-bound or exaggerating symptoms
Improvement in Functional Capacity of Neck | Immediate Intervention Group: Just before the intervention, immediately after (6 weeks), and 6 weeks post-intervention (12 weeks). Delayed Intervention Group: 6 weeks before the intervention, just before, and immediately after the intervention (6 weeks).
  Assessed using the the Neck Disability Index Questionnaire (NDI). Thise tool evaluates limitations in daily activities and the functional impact of cervical.
  The score ranges from 0 to 50, where higher scores indicate greater disability:
  0-4 (0-8%): No disability 5-14 (10-28%): Mild disability 15-24 (30-48%): Moderate disability 25-34 (50-68%): Severe disability 35-50 (70-100%): Complete disability
Reduction in Perceived Stress | Immediate Intervention Group: Just before the intervention, immediately after (6 weeks), and 6 weeks post-intervention (12 weeks). Delayed Intervention Group: 6 weeks before the intervention, just before, and immediately after the intervention (6 weeks).
  Measured using the Perceived Stress Scale (PSS), which quantifies participants' perceived stress levels over the last month by scoring their feelings and thoughts.
  The PSS ranges from 0 to 40, where higher scores indicate greater perceived stress. Scores between 0-13 suggest low stress, 14-26 indicate moderate stress, and 27-40 reflect high perceived stress.
Enhancement in Range of Motion | Immediate Intervention Group: Just before the intervention, immediately after (6 weeks), and 6 weeks post-intervention (12 weeks). Delayed Intervention Group: 6 weeks before the intervention, just before, and immediately after the intervention (6 weeks).
  Measured using a goniometer to determine improvements in cervical and lumbar spinal flexibility by quantifying the range of motion during specific movements.
Changes in Muscle Tone | Immediate Intervention Group: Just before the intervention, immediately after (6 weeks), and 6 weeks post-intervention (12 weeks). Delayed Intervention Group: 6 weeks before the intervention, just before, and immediately after the intervention (6 weeks).
  Evaluated using the Myoton device, which provides precise measurements of muscle tone, elasticity, and stiffness in the cervical and lumbar regions.
Improvement in Postural Alignment and Symmetry | Immediate Intervention Group: Just before the intervention, immediately after (6 weeks), and 6 weeks post-intervention (12 weeks). Delayed Intervention Group: 6 weeks before the intervention, just before, and immediately after the intervention (6 weeks).
  Assessed using the Motiphysio Scanner, which evaluates the alignment and symmetry of the spine and detects postural imbalances.
Improvement in Posture | Group 1: Baseline (just before the intervention), immediately after the intervention (6 weeks), and 6 weeks post-intervention (12 weeks after starting). Group 2: 6 weeks before the intervention, just before the intervention, and immediately after the int
  Measured using the Spinal Mouse technology, which captures detailed data on spinal curvature, segmental mobility, and overall spinal stability during various postures and movements. The units of measurement are degrees.

CONTACTS AND LOCATIONS:
Locations (1):
- Universidad San Jorge, Zaragoza, Zaragoza, Spain